CLINICAL TRIAL: NCT04137185
Title: Phase I/II Clinical Trial of Dose-tolerance, Pharmacokinetics and Iodine Uptake For Recombinant Human Thyroid Stimulating Hormone In Post-thyroidectomized Patients
Brief Title: Clinical Trial of Dose-tolerance, Pharmacokinetics and Iodine Uptake For rhTSH In Post-thyroidectomized Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGTSH001
Record Dates: First submitted 2019-09-20; First posted 2019-10-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — Thyrotropin Alfa; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhTSH (Experimental): Phase 1: 0.9mgx1d、0.9mgx2d、1.8mgx1d、1.8mgx2d, intramuscularly (IM) ; Phase 2: patients will be treated at the recommended dose for phase 2(RP2D).The RP2D will be determined by the Phase 1.
  Interventions: Drug: Recombinant Human Thyroid Stimulating Hormone for Injection

INTERVENTIONS:
Drug: Recombinant Human Thyroid Stimulating Hormone for Injection — rhTSH was dissolved in 1.2 mL of sterile water for injection to obtain a solution containing 0.9 mg/mL rhTSH.
  Other Names: rhTSH

SUMMARY:
Phase I/II Clinical Trial of Dose-tolerance, Pharmacokinetics and Iodine Uptake Effects For Recombinant Human Thyroid Stimulating Hormone In Post-thyroidectomized Patients

DETAILED DESCRIPTION:
This phase I/II study of rhTSH, To observe the safety and tolerability characteristics of different doses of rhTSH In Post-thyroidectomized Patients, and to observe the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of differentiated thyroid cancer, including papillary thyroid cancer (including papillary carcinoma follicular subtype), follicular thyroid cancer, and Hurthle cell thyroid cancer;
* Screening ages 18-75 (including 18 Age and 75 years old, male or female;
* Weight 45kg-80kg (including 45kg and 80kg, limited to the dose escalation test);
* Complete thyroidectomy or near total resection, and plan to start 131I diagnosis or ablation Patients
* Serum TSH ≤ 0.5 mU/L;
* Women of childbearing age are HCG-negative and must continue contraception until more than 3 months after the end of the trial;
* Subjects (including partners) from 2 weeks prior to dosing to the last study drug There is no pregnancy plan within 3 months after the drug and voluntary effective contraceptive measures are taken. For specific contraceptive measures, see Appendix 3;
* Normal ECG. Intermittent atrial premature beats, supraventricular tachycardia (SVT) or supraventricular block-independent PR interval abnormalities, right bundle branch block, mild sinus bradycardia (asymptomatic, and no treatment required) Can be grouped;
* Low iodine diet before enrollment for more than 4 weeks;
* Patients are voluntarily enrolled, and written informed consent forms can be used for treatment and visits as required by the program.

Exclusion Criteria:

* Patients who are not eligible for THST withdrawal due to pituitary disease or other diseases;
* Patients not eligible for 131I diagnosis or treatment;
* Any significant clinical and laboratory abnormalities (eg, severe cardiopulmonary disease, hepatic insufficiency, renal function) Incomplete, congestive heart failure, advanced lung disease or advanced cardiovascular and cerebrovascular disease, active infection);
* Hypertensive patients who cannot be reduced to the following range due to medical treatment (systolic blood pressure <140 mmHg, diastolic blood pressure <90 mmHg);
* Patients who have used any water-soluble radiographic contrast agent intravenously within 4 weeks before administration;
* Patients who underwent intrathecal iodine angiography or gallbladder iodine imaging within 3 months prior to administration;
* taken/eaten within 4 weeks prior to administration Drugs/foods that affect iodine uptake or metabolism, such as multivitamins, glucocorticoids, diuretics, lithium, thiouracil, tazobactam, algae, iodine (except thyroid hormone replacement therapy);
* before administration Stroke, unstable angina (CCS class II or higher), atrial fibrillation or medication (within beta blocker or digoxin) within 6 months Patients with a history of arrhythmia;
* pregnant or lactating women;
* a history of drug use and/or alcohol abuse within 3 months prior to dosing;
* patients who are allergic to rhTSH and its excipients;
* patients with positive infection-related tests : Includes hepatitis C and AIDS;
* Participated in any drug or medical device clinical trial within 1 month prior to the trial;
* Those who were unable to participate in the trial as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
MTD | up to 7 days
  the maximum tolerated dose

SECONDARY OUTCOMES:
Cmax | up to 5 days
  maximum serum thyrotropin concentrations
AUC | up to 5 days
  area under curve of serum thyrotropin concentration
Serum Tg | up to 7 days
  serum Tg levels
radioiodine uptake | up to 8 weeks
  whole body radioiodine imaging after rhTSH administration and after thyroid hormone withdrawal
adverse event | up to 8 weeks
  classification and degree of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China